CLINICAL TRIAL: NCT02323841
Title: Feasibility Study: Conservative Treatment in Cervical Cancer FIGO Stage IB1-IIA1 > 2cm
Brief Title: Feasibility Study: Conservative Treatment in Cervical Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Feasibility Study: Conservative Treatment in Cervical Cancer FIGO Stage IB1-IIA1 > 2cm, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 12650/13
Record Dates: First submitted 2014-04-08; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-02

CONDITIONS: Stage IB1 Cervical Cancer
Keywords: cervical cancer; neoadjuvant chemotherapy; Adverse Effects
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- conservative treatment in cervix cancer (Experimental): we performed conservative treatment cervix cancer patients with IB FIGO stage without pelvic involvement
  Interventions: Procedure: conservative treatment

INTERVENTIONS:
Procedure: conservative treatment — we performed pelvic lymphadenectomy before neoadjuvant chemotherapy and conization as conservative treatments

SUMMARY:
Currently conservative treatment for patients of childbearing affected by cervical cancer is reserved for women with FIGO stage IA2 - IB1 with tumor size less than 2 cm . The trachelectomy and the cone biopsy with pelvic lymphadenectomy are the choice for these patients wishing to preserve their reproductive function.

In this context , recently literature show the results about the use of neo-adjuvant chemotherapy about the reduction of tumor volume and therefore the magnitude of the subsequent surgical treatment (including patients with tumors larger than 2 cm ). So it becomes crucial a prospective analysis on the possibility to include in this type of treatment patients with stage IB1 and IIA1 with tumor size greater than 2 cm ( up to 4 cm ) .

The current study , in fact , would like to do a prospective evaluation on the advantages of neo-adjuvant chemotherapy in the possibility of broadening the inclusion criteria to conservative treatment in women , suffering from cervical cancer, stage IB1 and IIA1 ( with tumor volume between 2 and 4 cm) and wishing to preserve their reproductive function.

DETAILED DESCRIPTION:
The investigators would like to be conservative in young patients affected by early stage cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cervical cancer or adenocarcinoma in FIGO stage IB1-IIA, tumor volume between > 2 and ≤ 4 cm (instrumental evaluation).
* Informed consensus
* Childbearing
* Fertility (through US and ormonal withdrawal pre - e post neoadjuvant chemotherapy
* ASA (American Society of Anesthesiologist) Class < 2

Exclusion Criteria:

* ongoing pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | 3 years
  time of pregnancy. Case of miscarriage, pre-term delivery or full term delivery.

SECONDARY OUTCOMES:
disease free survival | 5 years
  time of disease free surviva
Overall survival | 5 years
  Time to the last follow up/death

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, PhD, Study Chair — Catholic University of Sacred Heart
Locations (1):
- Giovanni Scambia, Rome, Italy, Italy

REFERENCES:
- [Derived] Russo L, Gui B, Micco M, Panico C, De Vincenzo R, Fanfani F, Scambia G, Manfredi R. The role of MRI in cervical cancer > 2 cm (FIGO stage IB2-IIA1) conservatively treated with neoadjuvant chemotherapy followed by conization: a pilot study. Radiol Med. 2021 Aug;126(8):1055-1063. doi: 10.1007/s11547-021-01377-1. Epub 2021 May 31. PMID 34060027
- [Derived] de Vincenzo R, Ricci C, Fanfani F, Gui B, Gallotta V, Fagotti A, Ferrandina G, Scambia G. Neoadjuvant chemotherapy followed by conization in stage IB2-IIA1 cervical cancer larger than 2 cm: a pilot study. Fertil Steril. 2021 Jan;115(1):148-156. doi: 10.1016/j.fertnstert.2020.07.006. Epub 2020 Oct 20. PMID 33092819